CLINICAL TRIAL: NCT04086784
Title: 3D-printed Porous Titanium Alloy Cages Versus PEEK Cages: Pedicle Screw Loosening Rate and Fusion Rate in Patients With Osteoporosis
Brief Title: 3D-printed Porous Titanium Alloy Cages Versus PEEK Cages in Patients With Osteoporosis
Acronym: 3DCOP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Li Weishi, Director of the orthopaedic department, Peking University Third Hospital
Other Study IDs: M2019270
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Osteoporosis; Degenerative Disc Disease; Degenerative Lumbar Spinal Stenosis; Degeneration Spine
Keywords: 3D-printed Porous Titanium Alloy cage;PEEK cage;Osteoporosis
MeSH Terms: conditions — Osteoporosis; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3D-printed Cage: Patients undergoing posterior lumbar interbody fusion with 3D-printed Porous Titanium Alloy Cages at the lowest fusion segment
- Peek Cage: Patients undergoing posterior lumbar interbody fusion with PEEK Cages at the lowest fusion segment

SUMMARY:
This is a prospective,observational single-center study. The osteoporotic patients requiring posterior lumbar interbody fusion(PLIF) with cages at the lowest fusion segment are prospectively enrolled and followed up. The patients undergoing PLIF with the 3D-printed porous titanium alloy cages are compared with those using PEEK cages. The hypothesis is that the use of 3D-printed porous titanium alloy cages can reduce the rate of pedicle screw loosening and increase the rate of lumbar fusion in osteoporotic patients.

DETAILED DESCRIPTION:
Pedicle screw fixation is a widely used technique for the surgical treatment of degenerative lumbar diseases, which can stabilize the spine before solid fusion and restore spinal balance. However, because of population aging and the high rate of osteoporosis in the elderly with lumbar degenerative diseases, the pedicle screw loosening has become a frequently reported complication. The bone-screw interface in osteoporotic spine is unstable, leading to reduced pull-out force and cut-out force. Most of the previous studies only focused on the methods used to directly strengthen the pedicle screws, few of them explored the feasibility of reducing the loosening rate by accelerating the lumbar fusion precess.

The 3D-printed porous titanium alloy cages have been proved to have advantages in speeding up and enhancing the lumbar fusion over conventional PEEK cages. Therefore, we hypothesize that patients undergoing PLIF with 3D-printed cages can achieve lumbar fusion earlier than those using PEEK cages, thus the 3D-printed cages can reduce the load on pedicle screws sooner than PEEK cages. Finally, the 3D-printed cages can reduce the loosening rate and increase the fusion rate.

The osteoporotic patients requiring posterior lumbar interbody fusion(PLIF) with cages at the lowest fusion segment are prospectively enrolled and followed up. The researchers will invite appropriate patients to participate in the study after their surgical plans are determined. General patients data are collected after informed consent, such as age, gender, weight, height, bone mineral density measured in T-scores and Hounsfield units, detailed surgical plans, and etc. They are followed up at 3, 6, 12, and 24 months according to our clinical routine, including lumbar x-ray and certain questions about the clinical outcomes. In addition, this study requires the patients to have lumbar CT scans when the fusion status is unclear in x-ray, especially for the 6 months follow-up.

The patients undergoing PLIF with the 3D-printed porous titanium alloy cages are compared with those using conventional PEEK cages. The primary endpoints are the loosening rate and fusion rate at 6 months follow-up. The secondary endpoints are the loosening rate and fusion rate at other time point of follow-up , and the clinical outcomes(ODI and VAS) at every follow-up.

ELIGIBILITY:
Inclusion Criteria:

* aged≥ 50 years old
* lumbar degenerative diseases requiring lumbar fusion with pedicle screw fixation, such as degenerative lumbar spinal stenosis, degenerative lumbar spondylolisthesis.
* no response to nonoperative treatment of at least 3 months
* osteoporosis diagnosed by any method for bone mineral density evaluation, such as DXA, QCT，or vertebral Hounsfield units
* the lowest instrumented vertebrae were at L5 or S1
* the surgical plan includes lumbar interbody fusion with cages at the lowest fusion level
* informed consent

Exclusion Criteria:

* the surgical plan includes any techniques used to strengthen the fixation,such as augmentation of the pedicle screw with bone cement
* no lumbar CT scans within 3 months before the surgery
* no dual energy x-ray absorptiometry within 6 months before the surgery
* spondylolysis
* allergic to metal
* history of lumbar fusion surgery
* cervical myelopathy，thoracic spinal stenosis, motor neuron disease,tuberculosis of spine,spinal tumor

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the orthopaedic department of the Peking University Third Hospital, the osteoporotic in-patients requiring lumbar fusion with pedicle screw for lumbar degenerative diseases are invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pedicle screw loosening rate at the lowest instrumented vertebrae | 6 months
  The presence of radiolucent zones of ≥ 1mm thick around the pedicle screws, broken screws, or obvious screw back-out and cut-out on x-ray images.
Fusion rate at the lowest fusion level | 6 months
  The presence of continuous fusion mass at bone graft site in CT scans and less than 3 degree of intervertebral mobility on lateral flextion-extension x-ray images.

SECONDARY OUTCOMES:
Pedicle screw loosening rate at the lowest instrumented vertebrae | 3 months;12 months; 24 months
  The presence of radiolucent zones of ≥ 1mm thick around the pedicle screws, broken screws, or obvious screw back-out and cut-out on x-ray images.
Fusion rate at the lowest fusion level | 3 months;12 months; 24 months
  The presence of continuous fusion mass at bone graft site in CT scans and less than 3 degree of intervertebral mobility on lateral flextion-extension x-ray images.
Disability | 3 months; 6 months;12 months; 24 months
  The Oswestry Disability Index (ODI) (0-100) is used to assess disability.
Back pain | 3 months; 6 months;12 months; 24 months
  The Visual Analog Scale (VAS 0-10) is used the evaluate back pain.
Leg pain | 3 months; 6 months;12 months; 24 months
  The Visual Analog Scale (VAS 0-10) is used the evaluate leg pain.

CONTACTS AND LOCATIONS:
Overall Officials: Weishi Li, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will make the clinical study report available for half a year after the publication of the results of the study.
Supporting Information: CSR
Time Frame: The IPD will become available for half a year after the publication of the results of the study.
Access Criteria: The IPD is available to the readers of the journal in which our research is published. The corresponding author of the published papers will review the requests.

REFERENCES:
- [Background] Pannell WC, Savin DD, Scott TP, Wang JC, Daubs MD. Trends in the surgical treatment of lumbar spine disease in the United States. Spine J. 2015 Aug 1;15(8):1719-27. doi: 10.1016/j.spinee.2013.10.014. Epub 2013 Oct 31. PMID 24184652
- [Background] Amirouche F, Solitro GF, Magnan BP. Stability and Spine Pedicle Screws Fixation Strength-A Comparative Study of Bone Density and Insertion Angle. Spine Deform. 2016 Jul;4(4):261-267. doi: 10.1016/j.jspd.2015.12.008. Epub 2016 Jun 16. PMID 27927514
- [Background] Okuyama K, Abe E, Suzuki T, Tamura Y, Chiba M, Sato K. Influence of bone mineral density on pedicle screw fixation: a study of pedicle screw fixation augmenting posterior lumbar interbody fusion in elderly patients. Spine J. 2001 Nov-Dec;1(6):402-7. doi: 10.1016/s1529-9430(01)00078-x. PMID 14588296
- [Background] Bredow J, Boese CK, Werner CM, Siewe J, Lohrer L, Zarghooni K, Eysel P, Scheyerer MJ. Predictive validity of preoperative CT scans and the risk of pedicle screw loosening in spinal surgery. Arch Orthop Trauma Surg. 2016 Aug;136(8):1063-7. doi: 10.1007/s00402-016-2487-8. Epub 2016 Jun 16. PMID 27312862
- [Background] Chen P, Li Z, Hu Y. Prevalence of osteoporosis in China: a meta-analysis and systematic review. BMC Public Health. 2016 Oct 3;16(1):1039. doi: 10.1186/s12889-016-3712-7. PMID 27716144
- [Background] Galbusera F, Volkheimer D, Reitmaier S, Berger-Roscher N, Kienle A, Wilke HJ. Pedicle screw loosening: a clinically relevant complication? Eur Spine J. 2015 May;24(5):1005-16. doi: 10.1007/s00586-015-3768-6. Epub 2015 Jan 24. PMID 25616349
- [Background] Tokuhashi Y, Matsuzaki H, Oda H, Uei H. Clinical course and significance of the clear zone around the pedicle screws in the lumbar degenerative disease. Spine (Phila Pa 1976). 2008 Apr 15;33(8):903-8. doi: 10.1097/BRS.0b013e31816b1eff. PMID 18404111
- [Background] Bokov A, Bulkin A, Aleynik A, Kutlaeva M, Mlyavykh S. Pedicle Screws Loosening in Patients With Degenerative Diseases of the Lumbar Spine: Potential Risk Factors and Relative Contribution. Global Spine J. 2019 Feb;9(1):55-61. doi: 10.1177/2192568218772302. Epub 2018 May 24. PMID 30775209
- [Background] Goldstein CL, Brodke DS, Choma TJ. Surgical Management of Spinal Conditions in the Elderly Osteoporotic Spine. Neurosurgery. 2015 Oct;77 Suppl 4:S98-107. doi: 10.1227/NEU.0000000000000948. PMID 26378363
- [Background] Janssen I, Ryang YM, Gempt J, Bette S, Gerhardt J, Kirschke JS, Meyer B. Risk of cement leakage and pulmonary embolism by bone cement-augmented pedicle screw fixation of the thoracolumbar spine. Spine J. 2017 Jun;17(6):837-844. doi: 10.1016/j.spinee.2017.01.009. Epub 2017 Jan 17. PMID 28108403
- [Background] McGilvray KC, Easley J, Seim HB, Regan D, Berven SH, Hsu WK, Mroz TE, Puttlitz CM. Bony ingrowth potential of 3D-printed porous titanium alloy: a direct comparison of interbody cage materials in an in vivo ovine lumbar fusion model. Spine J. 2018 Jul;18(7):1250-1260. doi: 10.1016/j.spinee.2018.02.018. Epub 2018 Feb 26. PMID 29496624
- [Background] Li P, Jiang W, Yan J, Hu K, Han Z, Wang B, Zhao Y, Cui G, Wang Z, Mao K, Wang Y, Cui F. A novel 3D printed cage with microporous structure and in vivo fusion function. J Biomed Mater Res A. 2019 Jul;107(7):1386-1392. doi: 10.1002/jbm.a.36652. Epub 2019 Mar 18. PMID 30724479